CLINICAL TRIAL: NCT04738929
Title: Comparing Acute Effects of Extra Virgin Coconut Oil and Extra Virgin Olive Oil Consumption on Appetite and Food Intake in Normal Weight and Obese Male Subjects
Brief Title: Comparing EVCO and EVOO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Collaborators: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ziyaerokaymetin, Principal Investigator, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EVCO
Record Dates: First submitted 2021-01-20; First posted 2021-02-04 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Obesity; Appetitive Behavior
Keywords: Extra virgin coconut oil; medium chain fatty acids; extra virgin olive oil; obesity; peptide YY; resting metabolic rate.
MeSH Terms: conditions — Obesity; Appetitive Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal weight (Experimental): Normal weight subjects (BMI=18.5-25)
  Interventions: Other: Extra virgin coconut oil or extra virgin olive oil
- Obese (Experimental): Obese subjects (BMI=30-34.99)
  Interventions: Other: Extra virgin coconut oil or extra virgin olive oil

INTERVENTIONS:
Other: Extra virgin coconut oil or extra virgin olive oil — Subjects consumed standard breakfast meals containing "extra virgin coconut oil" or "extra virgin olive oil"

SUMMARY:
The aim of this study is to compare acute effects of consuming extra virgin coconut oil (EVCO) as a source of medium chain fatty acids and extra virgin olive oil (EVOO) as a source of long chain fatty acids in normal weight and obese subjects.

DETAILED DESCRIPTION:
Twenty male subjects (10 normal weight; 10 obese) consumed breakfast meals containing skimmed milk, fat-free white cheese, bread and EVCO (25 g) or EVOO (25 g). Visual analog scale evaluations, resting metabolic rate measurements and selected blood parameters analysis (glucose, triglyceride, insulin and plasma peptide YY) were performed before and after the test breakfast meals. In addition, energy intakes were evaluated by ad libitum lunch meal at 180 min.

ELIGIBILITY:
Inclusion Criteria:

* Metabolically healthy
* Aged 19-40 years
* Normal weight (BMI=18.5-24.9 kg/m²) and obese men (BMI=30-34.99 kg/m²)

Exclusion Criteria:

* smoking,
* alcohol consumption,
* weight gain/loss recently (> %5, in three months),
* any genetic and metabolic diseases,
* any food allergy/intolerance,
* any medication,
* restrained eating habits.

Ages: 19 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only male subjects were included to eliminate potential variations due to hormonal changes during menstrual cycles of female subjects.
Enrollment: 20 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2019-06-03 (Actual); Study Completion 2019-06-03 (Actual)

PRIMARY OUTCOMES:
Energy expenditure change | 0, 60, 120, 180 minutes
  kcal
Subjective appetite feelings change | 0, 30, 60, 120, 180 minutes
  visual analogue scales rating (0-10 cm)
glucose change | 0, 30, 60, 120, 180 minutes
  mg/dl
insulin change | 0, 30, 60, 120, 180 minutes
  mU/L
peptide YY change | 0, 30, 60, 120, 180 minutes
  pg/dl
triglycerides change | 0, 30, 60, 120, 180 minutes
  mg/dl
Ad libitum energy intake | 180 minute
  kcal

CONTACTS AND LOCATIONS:
Overall Officials: Ziya Erokay Metin, Dr., Principal Investigator — Ankara City Hospital Bilkent; Pelin Bilgiç, Assoc. Prof., Study Chair — Hacettepe University; Mercan Merve Tengilimoğlu Metin, Assis. Prof., Study Chair — Hacettepe University; Muzaffer Akkoca, Assoc. Prof., Study Chair — Saglik Bilimleri Universitesi
Locations (1):
- Presidency of Republic of Turkey Health Center, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Metin ZE, Bilgic P, Tengilimoglu Metin MM, Akkoca M. Comparing acute effects of extra virgin coconut oil and extra virgin olive oil consumption on appetite and food intake in normal-weight and obese male subjects. PLoS One. 2022 Sep 16;17(9):e0274663. doi: 10.1371/journal.pone.0274663. eCollection 2022. PMID 36112590